CLINICAL TRIAL: NCT01466088
Title: Double-Blind, Positive Comparator, Randomized, Parallel Study of Efficacy, Safety, and Tolerability of AZD3480 (TC-1734-226) as Monotherapy in Patients With Mild to Moderate Dementia of the Alzheimer's Type
Brief Title: Efficacy, Safety, & Tolerability of AZD3480 Patients With Mild to Moderate Dementia of the Alzheimer's Type (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-1734-226-CRD-006
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; AD; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Donepezil; ispronicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD3480 (Experimental)
  Interventions: Drug: AZD3480
- Donepezil (Active Comparator): Donepezil will be administered at 5 mg daily for 4 weeks and escalated to 10 mg daily for the remainder of the study.
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Subjects taking donepezil will take 1-2 capsules of 5 mg donepezil and a placebo for AZD3480 (to maintain blind) orally once a day.
  Other Names: Aricept
  Arms: Donepezil
Drug: AZD3480 — Subjects taking 30 mg AZD3480 will take one capsule of AZD3480 and two capsules of placebo for donepezil (to maintain blind) orally once a day.
  Other Names: TC-1734
  Arms: AZD3480

SUMMARY:
Alzheimer's disease is the most common form of dementia and is the fourth leading cause of death among people 65 years of age and older. The global prevalence of the disease will increase significantly as the population ages, unless preventative treatments can be identified and marketed. The present study seeks to evaluate AZD3480 (TC-1734) compared to an approved medication (donepezil) shown to improve cognition and function in patients with Alzheimer's disease.

DETAILED DESCRIPTION:
This is a double blind, positive comparator, randomized, multicenter, parallel group study to assess the efficacy, safety, and tolerability of AZD3480 as monotherapy in patients with mild to moderate dementia of the Alzheimer's type (AD). Approximately 300 subjects will be randomized and divided into 2 cohorts. Actual randomization was 293 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of AD per NINCDS-ADRDA criteria; mild to moderate severity as defined by Mini-Mental State Examination (MMSE) scores of 12 to 22.
2. AD diagnosed at least 12 months prior to Screening, and supported by brain imaging studies within 6 months prior to Screening.
3. Absence of vascular dementia both per AIRENS criteria and as defined by modified Hachinski ischemia score (HIS) of </= 4.
4. Presence of a caregiver with significant proportion of time in contact with subject and who will oversee administration of study drug during the trial
5. Able to complete test assessments and to sign informed consent with the help of a caregiver if needed

Exclusion Criteria:

1. Diagnosis or presence of other dementing illnesses
2. Use of mood stabilizers, antidepressants, anxiolytics, antipsychotics or hypnotics
3. Treatment within 1 month prior to Screening using cognition-affecting agents (e.g. CNS stimulants)
4. Tobacco user within 4 months prior to Screening
5. Use of smoking cessation therapy within 4 months prior to Screening
6. History within past 6 months of alcohol abuse or illicit drug abuse
7. Unable, even with caregiver assistance, to comply with study procedures in opinion of investigator
8. Myocardial infarction within the 12 months prior to Screening
9. Hypothyroidism, vitamin B12 or folic acid deficiency
10. Known systemic infection (HBV, HCV, HIV, TB)
11. Vascular dementia per NINDS-AIRENS criteria and as defined by a modified Hachinski ischemia score (HIS, Appendix 4) score of > 4 (i.e., vascular dementia is consistent with a modified HIS > 4).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog) | 52 weeks
Change from baseline in the Clinician Interview-Based Impression of Change plus carer interview [CIBIC-(+)] | 52 Weeks
  The CIBIC-(+) is a co-primary endpoint with the ADAS-Cog in the United States.
Change from baseline in the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | 52 Weeks
  The ADCS-ADL is the co-primary endpoint with the ADAS-Cog in Europe.

SECONDARY OUTCOMES:
Change from baseline in the Neuropsychiatric Inventory (NPI) | 52 Weeks
Change from baseline in the Mini-Mental State Examination (MMSE) | 52 Weeks
Change from baseline in the Alzheimer's Disease Related Quality of Life (ADRQL) | 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Tariot, MD, Principal Investigator — Banner Alzheimer Institute
Locations (33):
- United States (3):
  - Banner Alzheimer Institute, Phoenix, Arizona
  - Meridien Research, Brooksville, Florida
  - MD Clinical, Hallandale, Florida
- Czechia (8):
  - Policlinic, Choceň
  - BRAIN-SOULTHERAPY s.r.o., Kladno
  - Bialbi.s.r.o. Psychiatrické oddělení, Litoměřice
  - Psychiatricka Ambulance, Olomouc
  - Vojenska Nemocnice Psychiatricke oddeleni, Olomouc
  - Clintrial, Prague
  - PRAGTIS s.r.o., Prague
  - Psychosocialni centrum, Přerov
- Romania (5):
  - Crucea Alba - Dr. Oros si Asociatii - Societate Civila Medicala, Oradea
  - Spitalul de Psihiatrie Sibiu, Sibiu
  - Spitalul Clinic Judetean de Urgenta SIBIU, Sibiu
  - Spitalul Clinic Judetean de Urgenta, Clinica Psihiatrie, Timișoara
  - Spitalul Clinic Judetean de Urgenta, Clinica Neurologie 2, Timișoara
- Slovakia (4):
  - Neurologicka Ambulancia, s.r.o., Banská Bystrica
  - Univerzitna nemocnica Bratislava, Geronto-psychiatrické oddelenie, Bratislava
  - KONZILIUM s.r.o., Dubnica nad Váhom
  - Neurologická ambulancia, Krompachy
- Ukraine (13):
  - Dnipropetrovsk Regional Clinical Hospital, Dnipropetrovsk
  - Donetsk National Medical University of M. Gorky, Donetsk
  - Donetsk Regional Clinical Psychiatric Hospital, Donetsk
  - Crimean Republican Institution Psychoneurological Dispensary, Kerch
  - Central Clinical Hospital Ukrzaliznytsi, Kharkiv
  - Department of Age Physiology and Pathology of Nervous System; Institute of Gerontology NAMS, Kyiv
  - Lugansk Regional Clinical Psychoneurological Hospital, Luhansk
  - Lviv National Medical University named after Galytskyy, Lviv
  - Lviv Regional Clinical Psychiatric Hospital, Lviv
  - Odessa Regional Psychoneurology Dispensary, Odesa
  - Odessa Regional Psychiatric Hospital # 2, Oleksandrivka
  - Ukrainian Medical Stomatological Academy, Poltava
  - Department #3 of the Kherson Regional Psychiatric Hospital, Stepanovka